CLINICAL TRIAL: NCT01134029
Title: Planned CORR: Planned Care for Obesity and Risk Reduction
Acronym: Planned CORR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HL089444; UCSD# 2007-4401 (Other: UCSD)
Record Dates: First submitted 2010-02-10; First posted 2010-05-31 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Cardiovascular Risk Factors
Keywords: obesity; weight management and cardiovascular risk factors
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care (No Intervention): Control Group
- Stepped Care (Experimental): Intervention
  Interventions: Behavioral: Stepped Care

INTERVENTIONS:
Behavioral: Stepped Care — This group receives 2 years of a stepped care intervention including provider visits, health educator sessions, phone calls and mailings and availability of self management and group sessions, text messaging and a smoker's quit line.
  Other Names: Healthy Road to a Healthy Heart
  Arms: Stepped Care

SUMMARY:
The researchers propose a randomized controlled trial to evaluate how well an intervention, Planned Care for Obesity & Risk Reduction (Planned CORR), supports primary care treatment of obesity in adults with at least one cardiovascular risk factor (CVRF).

DETAILED DESCRIPTION:
The researchers propose a randomized controlled trial to evaluate how well an intervention, Planned Care for Obesity & Risk Reduction (Planned CORR), supports primary care treatment of obesity in adults with at least one cardiovascular risk factor (CVRF). We will assess how well it creates initial and sustained improvements in BMI and metabolic, anthropometric and behavioral outcomes in obese adults, age 25 to 70 who have one or more of the following CVRFs: hypertension, smoking or the metabolic syndrome. Planned CORR integrates intervention components based on behavior change theory with a delivery strategy based on the Chronic Care Model (Wagner et al, 2001; also called the "Planned Care Model") and is designed to incorporate intervention principles used successfully to treat obesity. Planned CORR is intended to be compatible with a variety of primary care settings including those with minimal resources to devote to patient education and where most obese adults receive their usual medical care. Study participants will be 380 women and men, age 25-70 who meet the entry criteria of obesity (Class I & II; BMI 30-45) plus one or more CVRFs. We anticipate that approximately 40% will be Hispanic and we will recruit an equal number of women and men and have powered the study to do analyses by gender. Planned CORR is a stepped care intervention that begins with computer-assisted assessment and tailored action planning, physician or nurse practitioner counseling, and an intensive "first step" of 4 months of lifestyle modification delivered via monthly in-person sessions and phone calls and weekly web or mail (based on preference) tutorials.CVRFs are managed concurrently according to recognized evidence-based protocols. Successive 4-month steps involve more, the same, or less intensive intervention depending on clinical response. The primary aim is to evaluate the effects at 12 & 24 months of Planned CORR on BMI when compared to enhanced usual care. Secondary aims will evaluate: CVRF outcomes; physiological, metabolic, behavioral, and psychosocial factors related to obesity and CVRFs; quality of life, depression and cost-effectiveness; and medical care quality, patient, provider & staff satisfaction, process measures relevant to implementation in primary care. Post study aims are to disseminate the knowledge gained from the intervention through conferences and publications, and to disseminate Planned CORR through proven channels of health care intervention dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 - 70
* English or Spanish Speaking
* Has transportation to get to follow-up appointments
* Has a functional and stable telephone number
* Lives in San Diego, maintains a permanent address, and plans on staying in San Diego for the next 2 years
* BMI of 30-45
* Have at least ONE of the following risk factors:

  * Hypertension
  * Smoking
  * Stabilized type II diabetes (Hemoglobin A1c Level <8.5);
  * Metabolic syndrome (defined as the presence of at least 3 of the following 5 factors: 1) elevated waist circumference: men: > 40 inches women: > 35 inches; 2) elevated triglycerides: >_150 mg/dL; 3) reduced HDL cholesterol: men < 40 mg/dL, women < 50 mg/dL; 4) elevated blood pressure: >130/85 mm.Hg; 5) Elevated fasting glucose (100-125 mg/dL).
* Able to participate in moderate physical activity

Exclusion Criteria:

* Has not had any form of bariatric/weight loss surgery (eg, gastric bypass, lap band) & does not intend to within 2 yrs.
* Does not have a history of substance abuse in the last 2 years (including amphetamines, opiates, and alcohol abuse) or other severe/unstable psychiatric disorder that would impair compliance with the study protocol (e.g. unstable depression, bipolar, schizophrenia).
* Is not pregnant or does not intend to become pregnant during the 2-year study period.
* Is not currently taking weight-altering medications (e.g. Sibutramine (Meridia), Orlistat (Xenical, Alli)), and has not taken them in at least 3 months.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the effects at 20 months of Planned CORR on BMI when compared to enhanced usual care. | 20 mo

SECONDARY OUTCOMES:
CVRF outcomes; physiological, metabolic, behavioral, and psychosocial factors related to obesity and CVRFs; quality of life, depression, cost-effectiveness; and medical care quality, patient, provider & staff satisfaction, and process measures. | 20 mo
CVRF outcomes; physiological, metabolic, behavioral, and psychosocial factors related to obesity and CVRFs; quality of life, depression, cost-effectiveness; and medical care quality, patient, provider & staff satisfaction, and process measures. | 8 months
CVRF outcomes; physiological, metabolic, behavioral, and psychosocial factors related to obesity and CVRFs; quality of life, depression, cost-effectiveness; and medical care quality, patient, provider & staff satisfaction, and process measures. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD - La Jolla Professional Building, La Jolla, California, United States

REFERENCES:
- [Derived] Liu J, Godino JG, Norman GJ, Hill L, Calfas K, Sallis JF, Arredondo E, Rock CL, Criqui M, Zhu SH, Griffiths K, Covin J, Dillon L, Patrick K. Planned care for obesity and cardiovascular risk reduction using a stepped-down approach: A randomized-controlled trial. Prev Med. 2018 Sep;114:223-231. doi: 10.1016/j.ypmed.2018.07.015. Epub 2018 Jul 25. PMID 30055199